CLINICAL TRIAL: NCT06261931
Title: Severity Over Time of Early Forms of Spondyloarthritis, a Prospective Observational Study.
Brief Title: Severity Over Time of Early Forms of Spondyloarthritis
Acronym: STAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6313
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Spondyloarthritis; Spondyloarthritis, Axial
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic assessment — patient with sponiloarthritis who comes to the clinic Hospital for clinical evaluation of disease. Assessment instrumental evaluation of the axial involvment t, with x-ray of the spine and pelvis every 5 years, and MRI of the spine and pelvis every 2 years.
Diagnostic Test: Diagnostic assessment — peripheral involvement, with joint ultrasound at baseline, at 3 months from the start of a new therapy, and therefore in the event of reactivation of the disease

SUMMARY:
Spondyloarthritis (SpA) is a group of chronic inflammatory pathologies whose progression over time is poorly defined, and in particular the clinical and instrumental elements that can predispose to a condition of disease severity are not completely known. It would be important to have an idea of what the predisposing factors are, possibly already at baseline, and possibly also at follow up, of severe disease, so as to be able to act early with more aggressive and targeted therapies on these patients, so as to achieve remission.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* Diagnosis of SpA confirmed by the rheumatologist with duration of symptoms <
* 2 years;
* Signature of the written informed consent to the study

Exclusion Criteria:

* Age < 18 years;
* Patients suffering from other rheumatic pathologies (even in overlap), or genetic diseases such as Marfan syndrome, Ehlers Danlos syndrome
* Any medical or psychiatric condition that in the judgment of the investigator would prevent the participant from complying with the protocol or completing the study according to the protocol.
* Refusal to sign the informed consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recent onset of SpA (duration of symptoms ≤2 years) and diagnosis made by the rheumatologist.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2044-02-28 (Estimated)

PRIMARY OUTCOMES:
spondyloarthritis severity | t0 baseline 3hours, t1 3 months 3hours,t2 6 months 3hours,t2 12months 3hours,every six months up to the tenth year
  evaluation of disease severity at 10 years in the entire study population

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided